CLINICAL TRIAL: NCT01144702
Title: Effectiveness of the Association Artesunate and Mefloquine in the Treatment of Uncomplicated Malaria by Plasmodium Falciparum, Juruá Valley, State of Acre, Brazil, 2009.
Brief Title: Effectiveness of the Association Artesunate and Mefloquine in the Treatment of Malaria by Plasmodium Falciparum
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Pan American Health Organization (Other); Ministry of Health, Brazil (Other Government); University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001/ASMQ/JURUA/2009
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Falciparum Malaria
Keywords: malaria; Plasmodium falciparum; artesunate and mefloquine combination (ASMQ); treatment; Juruá Valley; Brazil; multidrug resistance 1 gene of Plasmodium falciparum -Pfmdr1
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- artesunate & mefloquine combination (Experimental): ASMQ will be administered to individuals with uncomplicated malaria by P. falciparum according to the dose regimen for age and weight, standardized (Farmanguinhos, Ministry of Health). For patients in the range of 5 to <18kg (6 months to 5 years old), will be offered treatment in the pediatric presentation of Artesunate+Mefloquine 25 +50 mg (5 to <9 kg = 1 tablet once daily for 3 days, 9 to <18 kg = 2 tablets once daily for 3 days). To study subject aged 18 or more kilos (six years or more years old) will be given the combination of Artesunate + Mefloquine presentation ASMQ 100 +200 mg (18 to 29 kg = 1 tablet once daily for 3 days, 30 kg or more = 2 tablets once daily for 3 days). Clinically and biochemically monitoring will be done for 42 days.
  Interventions: Drug: artesunate & mefloquine combination

INTERVENTIONS:
Drug: artesunate & mefloquine combination — A therapeutic trial of a single arm for prospective evaluation of responses of individuals with uncomplicated malaria by P. falciparum treated with combination artesunate + mefloquine for three days and monitored clinically and biochemically for 42 days.
  Other Names: ASMQ

SUMMARY:
The purpose of this study was to evaluate the effectiveness of the fixed combination of artesunate+mefloquine in the treatment of uncomplicated malaria caused by Plasmodium falciparum in the municipality of Cruzeiro do Sul, Juruá Valley, Brazil, where it was being used as specific first-line drug.

DETAILED DESCRIPTION:
* Objectives: To evaluate the efficacy of the fixed combination of artesunate + mefloquine in the treatment of uncomplicated malaria caused by Plasmodium falciparum, in the county (municipality) of Cruzeiro do Sul, Juruá Valley, State of Acre (AC), Brazil, where it was being used as specific first-line drug.
* Selection Criteria : Persons aged between 6 months and 70 years with history of fever in the last 48 hours that had a confirmed diagnosis of mono-infection by Plasmodium falciparum (F or F+Fg) with parasitemia of 250 to 100000 parasites/μl and absence of signs of severe malaria, malnutrition or another severe disease. Pregnant women were not included.
* Intervention: Three days of supervised treatment with the fixed combination of artesunate+mefloquine (ASMQ-Farmanguinhos/Fiocruz) in accordance with the scheme recommended by the Ministry of Health, respecting four age and weight groups based on the target dose of each drug (artesunate -4 mg/kg/dose and 12 mg/kg of total dose, mefloquine- 8 mg/kg/dose and 24 mg/kg of total dose). Patients in the range of 5 to <18 kg (6 months to 5 years old) received the combination in pediatric presentation (ASMQ 25 + 50mg) and subjects with 18 kg or more (6 years or more years old) received the presentation ASMQ 100 + 200mg.
* Main Outcomes: The proportion of subjects who had experienced treatment failure during the following 42 days is used to estimate the effectiveness of the antimalarial combination in this study. Adverse events and speed of resolution of the clinical and infectious status are described. The phenotype of multidrug resistance (MDR) was investigated in the population of P. falciparum present in the subjects of the study.
* Methods: A therapeutic trial of a single "arm" for prospective evaluation of clinical and parasitological response of at least 100 individuals with uncomplicated malaria by P. falciparum treated with artesunate+mefloquine combination for three days and monitored for 42 days. The follow-up was done with assessments in the first four days and then once a week until the day 42. During the visits, subjects were submitted to an interview, clinical examination, temperature measurement and collection of venous (D0, D3 and D42) or capillar (all visits) blood samples for hemogram (D0, D3 and D42) and parasitological exam (all visits). The parasitological evaluation was done by microscopy (immediately with review later) and real time PCR (qPCR) in order to confirm the infecting specie of Plasmodium, to detect gametocytes and to measure the parasitemia (parasites/μl). ). The blood samples of D0 (before the treatment) was used to evaluate the phenotype of multidrug resistance (MDR) in the population of P. falciparum.
* Potential risks to participants: The action proposed does not add risks beyond those inherent to the treatment and course of illness, since the fixed combination artesunate + mefloquine was being used as the first line treatment of uncomplicated malaria caused by Plasmodium falciparum in the Valley Juruá since 2006 and still is recognized by the Ministry of Health as an alternative to the combination of artemether + lumefantrine in Brazil. If necessary, the study subjects could be admitted to the General Hospital Juruá seat of outpatient malaria. Medical and laboratory support was guaranteed free of charge to all study subjects and for all health problems that have been present during the follow-up.
* What the study adds to knowledge in public health? : This study offers a crucial knowledge to guide the development of policies to antimalarial drugs in endemic areas.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 6 months and 70 years old;
* Be with mono-infection confirmed laboratorial by P.falciparum;
* Having parasite count between 250/µl and 100000/µl;
* If female, not pregnant, confirmed by specific test;
* Being feverish or report having had fever (axillary temperature >37.5°C or 99,5°F) in last 48 hours;
* Be able to receive oral medication;
* Demonstrate interest and facility to meet the schedule of visits and monitoring for 42 days;
* Agree to participate in the study by signature (or parents) of Consent Term;
* Do not show evidence of severe malnutrition: underweight 60% of the weight-standard, below-average height for age indicating malnutrition in the past and weight-height below the average indicating dietary current deficiencies (WHO, 2006);
* Do not show danger signals to severe malaria. Note: We will be careful to include individuals who have used quinine or quinidine recently (three days before), because the risk of toxicity due to interaction with mefloquine.

Exclusion Criteria:

* Present after inclusion, danger signs/symptoms for severe malaria as recommended by the WHO;
* Present after inclusion, laboratory evidence of mixed infection with another species of Plasmodium;
* Having a diagnosis of other acute infectious disease that courses with fever, such as acute respiratory infection, common viruses of childhood diarrhea, etc;
* Having a diagnosis of chronic co morbidities or severe disease such as cirrhosis, chronic renal failure or heart failure;
* Have a history of hypersensitivity to the components of the combination ASMQ.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2010-11; Primary Completion 2013-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
treatment failure | 42 days
  The efficacy of the treatment will be based on clinical and parasitological evaluation of the participants, conducted in all follow-up visits during the 48 days. All individuals will be classified in: a) Early treatment failure b) Late Clinical Failure, Late Parasitological Failure and adequate clinical and parasitological response. As the parasitological cure is the endpoint of treatment of malaria, all individuals classified as treatment failure should be treated with the alternative scheme (quinine + doxycycline).

SECONDARY OUTCOMES:
Description of adverse events | 42 days
  Any sign or symptom that is not present in the clinical evaluation of D0 and focusing on subsequent evaluations, will be defined as adverse effects of the treatment. For this, a list of signs and symptoms should be questioned participants at all follow-up visits and adverse effects identified will be properly recorded. Depending on the intensity, these adverse effects should be treated according to medical advice. The subject of the study with more severe adverse effects will be referenced to a secondary or tertiary health care for the Juruá Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Simone L Andrade, PhD, Study Director — Oswaldo Cruz Institute, Oswaldo Cruz Foundation
Locations (2):
- Brazil (2):
  - Oswaldo Cruz Foundation, Rio de Janeiro, Rio de Janeiro
  - Institute of Biomedical Sciences, University of Sao Paulo, São Paulo, São Paulo

REFERENCES:
- [Derived] Ladeia-Andrade S, de Melo GN, de Souza-Lima Rde C, Salla LC, Bastos MS, Rodrigues PT, Luz Fd, Ferreira MU. No Clinical or Molecular Evidence of Plasmodium falciparum Resistance to Artesunate-Mefloquine in Northwestern Brazil. Am J Trop Med Hyg. 2016 Jul 6;95(1):148-54. doi: 10.4269/ajtmh.16-0017. Epub 2016 Apr 11. PMID 27068396